CLINICAL TRIAL: NCT05299164
Title: Liposomal Mitoxantrone Hydrochloride, Gemcitabine, Vinorelbine With or Without Rituximab (GVM±R) in Patients With Relapsed or Refractory Aggressive Non-Hodgkin's Lymphoma
Brief Title: GVM±R in Patients With Relapsed or Refractory Aggressive NHL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022003
Record Dates: First submitted 2022-03-10; First posted 2022-03-28 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma
Keywords: GVM±R; liposomal mitoxantrone hydrochloride
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: 3+3 dose-escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Liposomal mitoxantrone hydrochloride 16 mg/m^2 (with a caret included) (Experimental)
  Interventions: Drug: Liposomal Mitoxantrone Hydrochloride dose level 1
- Liposomal mitoxantrone hydrochloride 18 mg/m^2 (with a caret included) (Experimental)
  Interventions: Drug: Liposomal Mitoxantrone Hydrochloride dose level 2
- Liposomal mitoxantrone hydrochloride 20 mg/m^2 (with a caret included) (Experimental)
  Interventions: Drug: Liposomal Mitoxantrone Hydrochloride dose level 3
- Liposomal mitoxantrone hydrochloride 22 mg/m^2 (with a caret included) (Experimental)
  Interventions: Drug: Liposomal Mitoxantrone Hydrochloride dose level 4

INTERVENTIONS:
Drug: Liposomal Mitoxantrone Hydrochloride dose level 1 — Liposomal Mitoxantrone Hydrochloride 16 mg/m^2 (with a caret included) on day 1, every 3 weeks; Gemcitabine (800 mg/m^2) on day 1,8, every 3 weeks; Vinorelbine (25mg/m^2) on day 1,8, every 3 weeks; Rituximab (375mg/m^2) on day 1, every 3 weeks, only used in patients with CD20+ lymphoma;
  Arms: Liposomal mitoxantrone hydrochloride 16 mg/m^2 (with a caret included)
Drug: Liposomal Mitoxantrone Hydrochloride dose level 2 — Liposomal Mitoxantrone Hydrochloride 18 mg/m^2 (with a caret included) on day 1, every 3 weeks; Gemcitabine (800 mg/m^2) on day 1,8, every 3 weeks; Vinorelbine (25mg/m^2) on day 1,8, every 3 weeks; Rituximab (375mg/m^2) on day 1, every 3 weeks, only used in patients with CD20+ lymphoma;
  Arms: Liposomal mitoxantrone hydrochloride 18 mg/m^2 (with a caret included)
Drug: Liposomal Mitoxantrone Hydrochloride dose level 3 — Liposomal Mitoxantrone Hydrochloride 20 mg/m^2 (with a caret included) on day 1, every 3 weeks; Gemcitabine (800 mg/m^2) on day 1,8, every 3 weeks; Vinorelbine (25mg/m^2) on day 1,8, every 3 weeks; Rituximab (375mg/m^2) on day 1, every 3 weeks, only used in patients with CD20+ lymphoma;
  Arms: Liposomal mitoxantrone hydrochloride 20 mg/m^2 (with a caret included)
Drug: Liposomal Mitoxantrone Hydrochloride dose level 4 — Liposomal Mitoxantrone Hydrochloride 22 mg/m^2 (with a caret included) on day 1, every 3 weeks; Gemcitabine (800 mg/m^2) on day 1,8, every 3 weeks; Vinorelbine (25mg/m^2) on day 1,8, every 3 weeks; Rituximab (375mg/m^2) on day 1, every 3 weeks, only used in patients with CD20+ lymphoma;
  Arms: Liposomal mitoxantrone hydrochloride 22 mg/m^2 (with a caret included)

SUMMARY:
This is a prospective, dose-escalation clinical study to evaluate the safety and efficacy of GVM±R in patients with relapsed or refractory aggressive non-Hodgkin's lymphoma (NHL).

DETAILED DESCRIPTION:
This is a single-arm, single-center, dose-escalation clinical study to explore the maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride when combined with gemcitabine, vinorelbine and/or rituximab (GVM ± R) in patients with relapsed or refractory aggressive non-Hodgkin lymphoma (NHL). Liposomal mitoxantrone hydrochloride will be given on day 1 at four different doses (16 mg/m2, 18 mg/m2, 20 mg/m2,22 mg/m2) and be combined with gemcitabine, vinorelbine and/or rituximab (rituximab only in CD20+ lymphoma). The dose limited toxicity (DLT) will be evaluated after the first cycle of therapy. A maximum of 6 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign the informed consent
2. Age ≥18, ≤70years, no gender limitation
3. Expected survival ≥ 3 months;
4. Histologically confirmed diagnosis of aggressive NHL.
5. Subjects with relapsed or refractory NHL. Relapsed disease is defined as the disease relapsing after CR or PR, and the duration of prior response is more than 6 months. Refractory disease can be confirmed if any of the following conditions are met: 1) no PR or CR has been obtained after previous treatment; 2) CR / PR was achieved after prior therapy, but recurred within 6 months; 3) Recurrence after hematopoietic stem cell transplantation.
6. Subjects must have at least one evaluable or measurable lesion per lugano2014 criteria: for lymph node lesions, the length and diameter should be > 1.5cm; For non-lymph node lesions, the length and diameter should be > 1.0cm;
7. Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) : 0-1
8. The following baseline laboratory criteria are required: Absolute neutrophil count (ANC) ≥1.5×109/L, Platelet count (PLT) ≥75×109/ L, Hemoglobin(HB)≥ 80g/L, Total bilirubin (TBIL) ≤1.5X upper limit of normal (ULN), Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5X ULN, Serum creatinine (Scr) ≤1.5X ULN.

Exclusion Criteria:

1. The subject had previously received any of the following anti-tumor treatments:

   1. Subjects who have been treated with mitoxantrone or mitoxantrone liposomes;
   2. Previously received doxorubicin or other anthracycline treatment, and the total cumulative dose of doxorubicin was more than 360 mg/m2 (1 mg doxorubicin equivalent to 2 mg epirubicin);
   3. Subjects who received anti-tumor treatment (including chemotherapy, targeted therapy, glucocorticoid, traditional Chinese medicine with anti-tumor activity, etc.) or participated in other clinical trials and received trial drugs within 4 weeks before the first administration of the study drugs;
   4. Subjects who received autologous hematopoietic stem cell transplantation or allogeneic hematopoietic stem cell transplantation within 100 days of the first administration of study drugs;
2. Hypersensitivity to any study drug or its components;
3. Uncontrolled systemic diseases (such as active infection, uncontrolled hypertension, diabetes, etc.)
4. Heart function and disease meet one of the following conditions:

   1. Long QTc syndrome or QTc interval > 480 ms;
   2. Complete left bundle branch block, grade II or III atrioventricular block;
   3. Serious and uncontrolled arrhythmias requiring drug treatment;
   4. New York Heart Association grade ≥ III;
   5. Cardiac ejection fraction (LVEF)# 50%;
   6. A history of myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other arrhythmia requiring treatment, a history of clinically serious pericardial disease, or ECG evidence of acute ischemia or active conduction system abnormalities within 6 months before recruitment.

9. Hepatitis B and hepatitis C active infection (defined as hepatitis B virus surface antigen positive and hepatitis B virus DNA higher than 1x103 copy/mL; hepatitis C virus RNA high than 1x103 copy/mL) 10. Human immunodeficiency virus (HIV) infection (defined as HIV antibody positive) 11. Patients with other malignant tumors, except for effectively controlled non- melanoma skin basal cell carcinoma, breast/cervical carcinoma in situ or other tumors without treatment during the past 5 years. 12. Pregnant and lactating women and patients of childbearing age who are unwilling to take contraceptive measures; 13. Unsuitable subjects for this study determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2023-12-18 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | Through the last patient complete his DLT observation, assessed up to 21 days
  Maximum tolerated dose (MTD) of liposomal mitoxantrone hydrochloride in GVM±R

SECONDARY OUTCOMES:
Dose limited toxicities (DLTs) | Through the last patient complete his DLT observation, assessed up to 21 days
  adverse events (AE) defined as DLT events per protocol
The incidence rates of AE and SAE | up to 28 days after the last patient complete his study therapy
  AE or severe adverse events (SAE) occur since the first dose of therapy is given
Objective response rate (ORR) | up to 2 years
  Response is assessed according to the lugano criteria
Complete response rate (CRR) | : up to 2 years
  Response is assessed according to the lugano criteria
progression-free survival（PFS） | up to 2 years
  From the date of the first dose of therapy is given until disease progression, death or last follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Wei Liu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, CAMS & PUMC, Tianjin, Please Select, China

IPD SHARING:
Plan to Share IPD: No